CLINICAL TRIAL: NCT07050108
Title: Effect of Neurodynamic Moblization Versus Mulligan on Pain and Functional Abilities in Patients With Chronic Discogenic Sciatica
Acronym: DS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Asmaa ibrahim attia, principle investigator : Asmaa ibrahim Attia, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/004903
Record Dates: First submitted 2025-06-25; First posted 2025-07-03 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Sciatica; Discogenic Pain
Keywords: Neurodynamic Moblization; mulligan therapy; sciatica
MeSH Terms: conditions — Sciatica

STUDY DESIGN:
Intervention Model Description: neurodynamic ans mulligan
Who Masked: Outcomes Assessor
Masking Description: opaque sealed envelope
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- neurodynamic mobilization (Experimental): twenty two patients will receive neurodynamic mobilization and selected physical therapy program three times a week for four weeks
  Interventions: Other: neurodynamic mobilization; Other: selected physical therapy program
- Mulligan therapy (Experimental): twenty two patients will receive mulligan therapy and selected physical therapy program three times a week for four weeks
  Interventions: Other: mulligan therapy; Other: selected physical therapy program
- selected physical therapy program (Active Comparator): twenty two patients will selected physical therapy program three times a week for four weeks
  Interventions: Other: selected physical therapy program

INTERVENTIONS:
Other: neurodynamic mobilization — the patients will receive neurodynamic mobilization in the form of opening technique which include; static opening and dynamic opening. also, sliding and tensioning technique+ selected physical therapy program
  Arms: neurodynamic mobilization
Other: mulligan therapy — sustained natural apophyseal glide SNAGs are mobilisation techniques and are used as part of the Mulligan Concept+ selected physical therapy program The patient position is stitting on the edage of the plenth non weight bearing position. The therapist will stand behind the patient, the therapist will apply SNAG for 3 repetitions during the initial screening session,the patient will be asked to lean forwared while applying the technique .the therapist apply onle from fove to seven repetitions.patients who experienced no worsening or showed improvement of pain and ROM were considered good indication for the effectivness of treatment .
  Arms: Mulligan therapy
Other: selected physical therapy program — The program of therapeutic exercises consisted of upper and lower back exercises. Each exercise will repeat from ten to thirty times, three repetitions in three sets with rest one to two minutes between the sets. The repetition of each exercise vary according to the physical ability of each patient.
  Lower back strengthening exercises: From prone lying position, the patient will asked to raise one lower limb then the other then both lower limbs+ TENS and US

SUMMARY:
The purpose of the present study to compare between the effect of neurodynamic moblizaton and Mulligan SNAG's moblization on patients with chronic unilateral discogenic sciatica.

DETAILED DESCRIPTION:
Sciatica is a common problem in patients suffer from lumbar disc prolapse with an incidence of five cases per 1000 adults in developed countries . Sciatica causes significant disability. When applying neurodynamics, tension occurs in the nervous system, and pressure within the nerve increases due to the decrease of the cross-sectional area, and the axonal transport system lengthens the sciatic nerve after shortening because of the influence of the surrounding related structures and hamstring flexibility . After extention of the nerve and muscle, muscle performance is improved because of increases in the number of muscle fiber segments and cross-sectional area of muscle fibers.The majority of the research concerned with SNAG techniques has concentrated on the study of peripheral joints and the cervical region. Few studies have been concerned with the effects of SNAG on the lumbar spine. The rest of the available research was in the form of case reports or case series. Only 5 trials have investigated different effects of the SNAG technique when applied to the lumbar region. This study will improve the conservative treatment for sciatica and will decrease the cost of treatment and disability of the patient.

ELIGIBILITY:
Inclusion Criteria:

* All the patients diagnosed as lumbar radiculopathy (L5-S1) for at least six months. Diagnosis was confirmed by physical, neurological examination (motor assessment, sensory assessment, reflexes) and radiological assessment (CT or MRI).
* All patients has second grade of disc bulge which will detect from T2 axial view of MRI according to Fardon and Milette
* All patients has unilateral radiculopathy and pain in the distribution of scaitic nerve.
* The age of the patients will range from 35 to 50years . Their body mass index will range between( 22-25)

Exclusion Criteria:

* Bilateral and multilevel disc prolapse or bilateral radtadiating pain
* acute pain (pain less than three months).
* Presence of active infection in lumbar spine.
* Any other spinal deformities.
* Postoperative cases.
* Cauda equine lesion.
* Neoplasmic.
* Spinal stenosis.
* Mechanical low back pain.
* Failed back syndrome.

Ages: 35 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 66 (Estimated)
Dates: Start 2025-06-30 (Estimated); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
pressure pain threshold | up to four weeks
  ALgometer offer real-time visual & auditory feedback to control & monitor applied pressure rates to measure pressure pain threshold.
pain intensity | up to four weeks
  Sciatica Bothersomeness Index will be used to assess pain intensity. An index based on patients reporting of symptoms which reflects the troubled patient is going through with his sciatica symptoms. Items from the Sciatica Bothersomeness Index (0 = none to 6 = extremely) were used to establish values for paresthesia, weakness and leg pain.

SECONDARY OUTCOMES:
Range of motion assessment of straight leg raise | up to four weeks
  A unilevel inclinometer will be used to assess the straight leg raise (SLR) test. From supine lying position on a flat plinth towards the side of the examiner, with the neck in a neutral position. The examiner places one hand under the Achilles tendon and the other hand held the inclinometer. The inclinometer must be held in a vertical position during the SLR test by the examiner's hand between the index and the middle fingers and center of inclinometer will be positioned on the lower third of tibia. The leg will be lifted perpendicular to the point at which the patient expressed the perception of pain and the therapist will prevente any knee flexion. The angle of hip flexion during SLR will be measured
disability | up to four weeks
  Roland-Morris Disability Questionnaire will be used to assess disability.The RMQ is a 24-item patient-reported outcome measure that inquires about pain-related disability resulting from LBP and discogenic sciatica .total RMQ score ranging from 0 to 24; higher scores represent higher levels of pain-related disability